CLINICAL TRIAL: NCT02299765
Title: A Randomized, Open-label, Multiple-centre Study of Intercalating and Maintenance Gefitinib in Combination With Chemotherapy for Advanced NSCLC With EGFR Mutation Positive
Brief Title: Intercalating and Maintenance Gefitinib in Combination With Chemotherapy for Advanced EGFR-mutant NSCLC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the research data is not statistically significant
Sponsor: Sichuan University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, You Lu, Chief Physician, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSIRES0109
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic; EGFR Activating Mutation
Keywords: Advanced Non-small Cell Lung Cancer (NSCLC); EGFR Mutation; gefitinib; chemotherapy
MeSH Terms: interventions — Gefitinib; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Four cycles gemcitabine(d1,8 ) + carboplatin (d1) + gefitinib (15-25), gefitinib 250mg/d from d15 of last cycle until disease progression.
  Gemcitabine=1000mg/m2;Carboplatin 5×AUC ; One cycle is 28 days
  Interventions: Drug: Gefitinib; Drug: gemcitabine; Drug: carboplatin
- Arm B (Active Comparator): Gefitinib 250mg/d until disease progression
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — patients in arm A will be given gefitinib as target therapy
  Other Names: Iressa
Drug: gemcitabine — patients in arm A will be given gemcitabine chemotherapy
  Other Names: Gemza
  Arms: Arm A
Drug: carboplatin — patients in arm A will be given carboplatin chemotherapy
  Other Names: Carboplatin Injection
  Arms: Arm A

SUMMARY:
Study Title:

Intercalating and maintenance Gefitinib in combination with chemotherapy (gemcitabine plus carboplatin) as first-line treatment for patients with advanced EGFR mutation-positive non-small cell lung cancer: A randomized, open-label, multiple-centre study.

Target population-Treatment naive EGFR mutant-positive advanced NSCLC patients.

Study Objectives - Primary Study Objective: To investigate whether intercalating and maintenance Gefitinib in combination with chemotherapy improve the Progression-Free Survival (PFS) vs. Gefitinib alone in advanced NSCLC with EGFR activating mutation.

- Secondary Study Objective： To evaluate whether intercalating and maintenance Gefitinib in combination with chemotherapy improve the Objective Response Rate (ORR), Disease control rate (DCR), Overall survival (OS), 2-year OS rate, QOL vs. Gefitinib alone.

Evaluation the safety of Intercalating and Maintenance Gefitinib in combination with chemotherapy.

- Exploratory objective: PFS of arm A vs. PFS 1 + PFS 2 of arm B Dynamic biomarker analysis using blood sample

a: The PFS 1 of arm B is the time from randomization to disease progression of 1st-line therapy or death from any cause, whichever occurs first. The PFS 2 of arm B is the time from the time of PFS 1 to disease progression of 2nd-line therapy or death from any cause, whichever occurs first.

Study Design-Prospective, open-label, randomized, multi-center study.

DETAILED DESCRIPTION:
Study Design:

It is a two-arm, prospective, randomized, open-label, multi-center study. The study will be conducted at 5 study sites in China. West China Hospital serves as the lead site for the study. A total of 146 treatments naive EGFR mutant positive advanced NSCLC patients are planned to be enrolled into this study.

There are four periods in this study: baseline period (≤28days),main phase of treatment (Week 0-Week 16 or until disease progression),post-treatment period and follow-up until about 24 months after the last patients enrolment.

1. Baseline period: Subject will be enrolled in the study after signing informed consent form (ICF). Investigator will record patient-reported outcome, demographic data and medical history, collect the histological or cytological samples for genetic testing, conduct laboratory examination and perform imaging examination and so on. Notes: The time of imagination is effective within 4 weeks before treatment. The result of haematology, biochemistry and physical examination is effective within 7 days before treatment. Collecting blood one time at screening period (The SOP of blood collection, storage and transportation is in attachment 1).
2. Main phase of treatment: There are 8 visits during the main phase of treatment study. During the main phase of treatment, investigator conduct laboratory examination, perform imaging examination, assess the tumor status, and evaluate the patient-reported outcome and safety.

   Collecting blood one time every two cycles (The SOP of blood collection, storage and transportation is in attachment 1).
3. Post-treatment period:

   In the study group, investigators will conduct laboratory examination, perform imaging examination, assess the tumor status, and evaluate the patient-reported outcome and safety until disease progression every 8 weeks. And after disease progression investigators will enquire and record survival status of subjects every 8 weeks.

   In the control group, investigators will conduct laboratory examination, perform imaging examination, assess the tumor status, and evaluate the patient-reported outcome and safety until the first and the second disease progression every 8 weeks. In addition, the information conduct between first disease progression and second progression are optional, but should be collected if available. And after the second disease progression investigators will enquire and record survival status of subjects every 8 weeks.

   Collecting blood one time every 8 weeks until progress (for control group it will be until the first progress)
4. Follow-up period:

It will last until about 24 months after the last patients' enrolment. Accesses histological or cytological samples for EGFR testing and related drug resistant gene testing are required. In addition, collection blood is optional, but should be collected if available. All the samples collected during his/her whole life treatment are transported to West China Hospital to store and will be used for further exploratory analysis later.

All results of CT/MRI need to be burned into compact disc (CD). This study will be the first study to compare the efficacy of intercalating and maintenance gefitinib in combination with chemotherapy to gefitinib alone as first-line treatment for patients with advanced EGFR activating mutation-positive non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study are required to meet the following inclusion criteria:

  1. Patients between 18 and 75 years of age.
  2. Patients with histologically or cytologically diagnosed NSCLC,or patients with recurrent advanced NSCLC after surgery.
  3. Harboring activating mutation of EGFR,only including an exon 19 deletion or an exon 21 point mutation.
  4. Has at least one measureable lesion by RECIST 1.1
  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  6. No prior systemic chemotherapy or targeted therapy for lung cancer before screening except neoadjuvant or adjuvant patients.
  7. Adequate organ function, including the following:

     Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1.5 × 109/L,platelets ≥100 × 109/L,and hemoglobin ≥9 g/dL.

     Hepatic: bilirubin ≤1.5 times the upper limit of normal (× ULN),alkaline phosphatase (AP),aspartate transaminase (AST),and alanine transaminase (ALT) ≤3.0 × ULN (AP,AST and ALT ≤5 × ULN is acceptable if the liver has tumor involvement).

     Renal: calculated creatinine clearance (CrCl) ≥45 mL/minute based on the standard Cockcroft and Gault formula.
  8. Prior radiation therapy allowed to <25% of the bone marrow. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study enrolment.
  9. Signed informed consent document on file.
  10. Estimated life expectancy of ≥12 weeks.
  11. Patient compliance and geographic proximity that allow adequate follow up.

      Exclusion Criteria:
* Subjects meeting any of the following exclusion criteria are not to be enrolled in the study.

  1. Known severe hypersensitivity to gefitinib.
  2. Known brain metastasis unless asymptomatic brain metastasis(without neurotic symptoms and sign) and treated with surgery and/or radiation and stable without steroid treatment for at least 2 weeks prior to the first dose of study medication.
  3. Pleural effusion or pericardiac effusion that cannot be controlled by drainage or other procedures.
  4. Previous treatment with agents targeting the HER axis.
  5. Previous systemic antitumour treatment.
  6. The last regimen of neoadjuvant or adjuvant treatment for non-metastatic disease within 12 months of study treatment.
  7. EGFR Resistance mutation (+).
  8. Surgery undertaken less than 4 weeks before the study.
  9. Inability to comply with protocol or study procedures.
  10. A serious concomitant systemic disorder that,in the opinion of the investigator，would compromise the patient's ability to complete the study.
  11. A serious cardiac condition,such as myocardial infarction within 6 months,angina,or heart disease.
  12. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment.
  13. Past medical history of Interstitial Lung Disease(ILD),drug induced interstitial disease,radiation pneumonitis which required steroid treatment,or any evidence of clinically active ILD.
  14. Pre-existing idiopathic pulmonary fibrosis evidence by CT scan at baseline.
  15. Unwillingness to use contraception during the study, women who were pregnant or lactating.
  16. Being or planing to participate in other studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival - PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to average 10 months

SECONDARY OUTCOMES:
Objective Response Rate - ORR | at day 42 of treatment
Overall Survival - OS | the time from randomization to death from any cause,assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Study Director — Department of Thoracic Oncology, Cancer center, West China Hospital, Sichuan University
Locations (1):
- China West Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Han JY, Park K, Kim SW, Lee DH, Kim HY, Kim HT, Ahn MJ, Yun T, Ahn JS, Suh C, Lee JS, Yoon SJ, Han JH, Lee JW, Jo SJ, Lee JS. First-SIGNAL: first-line single-agent iressa versus gemcitabine and cisplatin trial in never-smokers with adenocarcinoma of the lung. J Clin Oncol. 2012 Apr 1;30(10):1122-8. doi: 10.1200/JCO.2011.36.8456. Epub 2012 Feb 27. PMID 22370314
- [Background] Giaccone G, Herbst RS, Manegold C, Scagliotti G, Rosell R, Miller V, Natale RB, Schiller JH, Von Pawel J, Pluzanska A, Gatzemeier U, Grous J, Ochs JS, Averbuch SD, Wolf MK, Rennie P, Fandi A, Johnson DH. Gefitinib in combination with gemcitabine and cisplatin in advanced non-small-cell lung cancer: a phase III trial--INTACT 1. J Clin Oncol. 2004 Mar 1;22(5):777-84. doi: 10.1200/JCO.2004.08.001. PMID 14990632
- [Background] Herbst RS, Giaccone G, Schiller JH, Natale RB, Miller V, Manegold C, Scagliotti G, Rosell R, Oliff I, Reeves JA, Wolf MK, Krebs AD, Averbuch SD, Ochs JS, Grous J, Fandi A, Johnson DH. Gefitinib in combination with paclitaxel and carboplatin in advanced non-small-cell lung cancer: a phase III trial--INTACT 2. J Clin Oncol. 2004 Mar 1;22(5):785-94. doi: 10.1200/JCO.2004.07.215. PMID 14990633
- [Background] Herbst RS, Prager D, Hermann R, Fehrenbacher L, Johnson BE, Sandler A, Kris MG, Tran HT, Klein P, Li X, Ramies D, Johnson DH, Miller VA; TRIBUTE Investigator Group. TRIBUTE: a phase III trial of erlotinib hydrochloride (OSI-774) combined with carboplatin and paclitaxel chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5892-9. doi: 10.1200/JCO.2005.02.840. Epub 2005 Jul 25. PMID 16043829
- [Background] Gatzemeier U, Pluzanska A, Szczesna A, Kaukel E, Roubec J, De Rosa F, Milanowski J, Karnicka-Mlodkowski H, Pesek M, Serwatowski P, Ramlau R, Janaskova T, Vansteenkiste J, Strausz J, Manikhas GM, Von Pawel J. Phase III study of erlotinib in combination with cisplatin and gemcitabine in advanced non-small-cell lung cancer: the Tarceva Lung Cancer Investigation Trial. J Clin Oncol. 2007 Apr 20;25(12):1545-52. doi: 10.1200/JCO.2005.05.1474. PMID 17442998
- [Background] Li T, Ling YH, Goldman ID, Perez-Soler R. Schedule-dependent cytotoxic synergism of pemetrexed and erlotinib in human non-small cell lung cancer cells. Clin Cancer Res. 2007 Jun 1;13(11):3413-22. doi: 10.1158/1078-0432.CCR-06-2923. PMID 17545550
- [Background] Cheng H, An SJ, Zhang XC, Dong S, Zhang YF, Chen ZH, Chen HJ, Guo AL, Lin QX, Wu YL. In vitro sequence-dependent synergism between paclitaxel and gefitinib in human lung cancer cell lines. Cancer Chemother Pharmacol. 2011 Mar;67(3):637-46. doi: 10.1007/s00280-010-1347-4. Epub 2010 May 22. PMID 20495920
- [Background] Piperdi B, Ling Y-H, Kroog G, et al. Schedule-dependent interaction between epidermal growth factor inhibitors (EGFRI) and G2/M blocking chemotherapeutic agents (G2/Mb) on human NSCLC cell lines in vitro [J]. J Clin Oncol, 2004; 22: 7028.
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Background] Wu YL, Lee JS, Thongprasert S, Yu CJ, Zhang L, Ladrera G, Srimuninnimit V, Sriuranpong V, Sandoval-Tan J, Zhu Y, Liao M, Zhou C, Pan H, Lee V, Chen YM, Sun Y, Margono B, Fuerte F, Chang GC, Seetalarom K, Wang J, Cheng A, Syahruddin E, Qian X, Ho J, Kurnianda J, Liu HE, Jin K, Truman M, Bara I, Mok T. Intercalated combination of chemotherapy and erlotinib for patients with advanced stage non-small-cell lung cancer (FASTACT-2): a randomised, double-blind trial. Lancet Oncol. 2013 Jul;14(8):777-86. doi: 10.1016/S1470-2045(13)70254-7. Epub 2013 Jun 17. PMID 23782814
- [Background] Yoshimura1 N, Matsuura1 K, Mitsuoka1 S, et al. Gefitinib(G) and pemetrexed（PEM）as a first line treatment in patients with EGFR mutation advanced non-small-cell cancer(NSCLC): a phase II study. ESMO 2012,1258p.
- [Background] Kanda S, Ohe Y, Horinouchi H, et al. Phase II study of gefitinib and inserted cisplatin plus docetaxel as a first-line treatment for advanced non-small cell lung cancer harboring an epidermal growth factor receptor activating mutation. ASCO Abstract, 2013,8064.
- [Background] Choi YJ, Kim SW, Lee DH, et al.Paclitaxel/carboplatin (PC) intercalated with gefitinib or paclitaxel/carboplatin (PC) for advanced non-small cell lung cancer (NSCLC) in selected population who were smoker or wild-type EGFR: Randomized phase II study. ASCO Abstract, 2013, e19079.
- [Background] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771
- [Background] Zhang L, Ma S, Song X, Han B, Cheng Y, Huang C, Yang S, Liu X, Liu Y, Lu S, Wang J, Zhang S, Zhou C, Zhang X, Hayashi N, Wang M; INFORM investigators. Gefitinib versus placebo as maintenance therapy in patients with locally advanced or metastatic non-small-cell lung cancer (INFORM; C-TONG 0804): a multicentre, double-blind randomised phase 3 trial. Lancet Oncol. 2012 May;13(5):466-75. doi: 10.1016/S1470-2045(12)70117-1. Epub 2012 Apr 17. PMID 22512843
- [Background] Cataldo VD, Gibbons DL, Perez-Soler R, Quintas-Cardama A. Treatment of non-small-cell lung cancer with erlotinib or gefitinib. N Engl J Med. 2011 Mar 10;364(10):947-55. doi: 10.1056/NEJMct0807960. PMID 21388312
- [Background] Kuo LC, Lin PC, Wang KF, Yuan MK, Chang SC. Successful treatment of gefitinib-induced acute interstitial pneumonitis with high-dose corticosteroid: a case report and literature review. Med Oncol. 2011 Mar;28(1):79-82. doi: 10.1007/s12032-010-9424-4. Epub 2010 Jan 20. PMID 20087691
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774